CLINICAL TRIAL: NCT02725827
Title: Randomized Controlled Trial Comparing Hyaluronan-enriched Embryo Transfer Medium Versus Control for Frozen-thawed Embryo Transfer
Brief Title: Hyaluronan-enriched Embryo Transfer Medium for Frozen-thawed Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Dr. YUNG Shuk Fei Sofie, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 16-158
Record Dates: First submitted 2016-03-23; First posted 2016-04-01 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: In Vitro Fertilization; Subfertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- HA group (Active Comparator): One the day of frozen-thawed embryo transfer, frozen embryos will be thawed and incubated for at least 10 minutes in embryo transfer medium. For women allocated to the HA group, EmbryoGlue (Vitrolife), a hyaluronan-enriched embryo transfer medium, will be used as embryo transfer medium. EmbryoGlue contains a higher concentration of hyaluronan than the control medium.
  Interventions: Other: EmbryoGlue (Vitrolife)
- Control group (Active Comparator): For women allocated to the control group, the usual transfer medium used in the study centers will be used and will serve as control. The main difference between the two media is that EmbryoGlue contains a higher concentration of HA.
  Interventions: Other: Control medium

INTERVENTIONS:
Other: EmbryoGlue (Vitrolife) — A hyaluronan-enriched embryo transfer medium
  Arms: HA group
Other: Control medium — The usual embryo transfer medium used in the study centres.
  Arms: Control group

SUMMARY:
This is a randomized-controlled trial evaluating the effect of the use of hyaluronan (HA)-enriched embryo transfer medium on the live birth rate in women undergoing frozen-thawed embryo transfer. For half of the women, hyaluronan-enriched medium will be used as embryo transfer medium. For the other half of women, a control will be used.

DETAILED DESCRIPTION:
Women being scheduled for FET will be assessed for eligibility. Eligible women will be recruited for the study and each woman will only be included in the study with one FET cycle. Informed written consent will be obtained. Their baseline characteristics will be collected.

Women with regular ovulatory cycles will undergo the standard procedures of blood taking to identify the day of luteinizing hormone (LH) surge. Women with irregular cycles will either receive clomiphene or letrozole followed by detection of the LH surge, or undergo hormone replacement therapy (HRT) cycle with oral oestradiol 6 mg daily for 14 days for endometrial priming followed by the addition of vaginal micronized progesterone 100 mg three times daily. HRT cycle may also be used for scheduling purposes.

Embryo transfer will be performed 3 or 4 days (for cleavage-stage embryos) or 6 or 7 days (for blastocysts) after the LH surge. For women in HRT cycles, FET will be scheduled on the 4th or 5th day (for cleavage-stage embryos) or the 7th or 8th day (for blastocysts) of starting vaginal progesterone. They will continue oral oestradiol and vaginal progesterone after FET up to 12 weeks of gestation.

Randomization:

One day before scheduled FET, recruited women will be randomized into one of the following two groups: (1) HA group and (2) control group according to a computer-generated randomization list prepared by a designated research nurse.

One the day of FET, frozen embryos or blastocysts will be thawed and incubated for at least 10 minutes in embryo transfer medium. For women allocated to the HA group, EmbryoGlue (Vitrolife) will be used as embryo transfer medium, while in the control group the usual medium used in the study center will used. The main difference between the two media is that EmbryoGlue contains a higher concentration of HA.

The rest of the embryo transfer procedure will be the same as the usual practice.

Blinding:

The patient and the physicians performing the FET and involved in her care will not know the group allocation. Only the embryologist will know the group allocation, but they will not be involved in the patient care, the FET procedure and subsequent assessment.

Follow-up and data collection:

A urine pregnancy test is performed 18 days after the LH surge or starting vaginal progesterone. If the pregnancy test is positive, transvaginal ultrasound will be performed 2 weeks later to locate the pregnancy and fetal viability. Subsequent management will be the same as other women with early pregnancy. They will be referred for antenatal care when the pregnancy is on-going at 8 weeks.

Follow-up:

Written consent regarding retrieval of pregnancy and delivery data from both public and private sectors will be sought from the patient at the time of study. The obstetric outcomes will be traced from the electric patient record system if the patients deliver in Hospital Authority hospitals. A pre-formatted letter with replying address available will be given to the patient at the end of the study period and is to be filled by the private obstetrician and returned to us after delivery. If no reply letter is received 2-3 months after the expected date of confinement of the patient, a letter including patient's authorization will be sent to the corresponding private obstetrician to retrieve the information of the pregnancy outcomes. The outcome of the pregnancy (delivery, miscarriage), number of babies born, birth weights and obstetrics complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women panning to replacing early cleavage embryos or blastocysts after thawing.

Exclusion Criteria:

* Frozen early cleavage embryos thawed and cultured to blastocysts prior to transfer as requested by the patient
* Preimplantation genetic diagnosis treatment
* Use of donor oocytes or donor embryos
* Endometrial thickness <8mm on the day of the luteinizing hormone surge or after two weeks of estrogen in hormonal replacement cycles
* Hydrosalpinx shown on pelvic scanning and not surgically treated

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Live-birth rate per embryo transfer procedure | 1 year

SECONDARY OUTCOMES:
pregnancy rate | 4 weeks
  positive urine pregnancy test
clinical pregnancy rate | 4 weeks
  presence of intrauterine gestational sac on ultrasound
implantation rate | 8 weeks
  number of gestational sacs per embryo transferred
on-going pregnancy rate | 8 weeks
  viable pregnancy beyond gestation 8 weeks
adverse events | 12 weeks
obstetric complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shuk Fei Sofie Yung, MBBS, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Kwong Wah Hospital, Hong Kong
  - Queen Mary Hospital, University of Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yung SSF, Lai SF, Lam MT, Lui EMW, Ko JKY, Li HWR, Wong JYY, Lau EYL, Yeung WSB, Ng EHY. Hyaluronic acid-enriched transfer medium for frozen embryo transfer: a randomized, double-blind, controlled trial. Fertil Steril. 2021 Oct;116(4):1001-1009. doi: 10.1016/j.fertnstert.2021.02.015. Epub 2021 Apr 9. PMID 33845988